CLINICAL TRIAL: NCT03883334
Title: Efecto de la Isoprinosina en Pacientes Con infección Por VIH y Carga Viral Entre > 50 y < 200 Copias/mL de la Unidad de atención de PVV Del Hospital Enrique Garcés en Quito, Ecuador Durante el año 2019.
Brief Title: Isoprinosine in HIV Patients With Viral Load > 50 y < 200 Copies/mL
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Universidad San Francisco de Quito (Other)
Responsible Party: Principal Investigator, Enrique Teran, Professor, Universidad San Francisco de Quito
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HUBI - 12522
Record Dates: First submitted 2019-02-07; First posted 2019-03-20 (Actual); Last update posted 2019-12-23 (Actual); Status verified 2019-12

CONDITIONS: HIV Infections
MeSH Terms: conditions — HIV Infections | interventions — Inosine Pranobex

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Immunomodulator group (Experimental): Metisoprinol 1 gr every 8 h per ten days during three months plus the combine antiretroviral therapy.
  Interventions: Drug: Metisoprinol
- Control group (No Intervention): combine antiretroviral therapy only

INTERVENTIONS:
Drug: Metisoprinol — Immunodulator
  Other Names: Isoprinosine
  Arms: Immunomodulator group

SUMMARY:
Virological failure is a complication of treatment in patients with HIV, and it can be as high as 42% to first line treatment or around 18% in second line treatment. The reasons behind this phenomenon are several, including adherence to treatment (self-patient) or those related to the drugs (kinetics, interactions) and the virus itself (resistance patterns). People living with HIV needs treatment for all their lives, another factor to facilitate virus resistance and poor adherence to treatment. For that reason, it is necessary to look for additional therapeutic options to minimize this problem, and the use of immunomodulatory drugs is an interesting topic now. Among those drugs, isoprinosine hs been reported not only improve the immune response, it also has the capability to inhibit the replication of RNA virus. Then, we propose an open label clinical trial to evaluate the effect of isoprinosine in HIV patients with a virological load between 50 and 200 copies/ml.

ELIGIBILITY:
Inclusion Criteria:

* Older than 18 years old.
* Patients with a viral load (RNA of VIH) between > 50 and < 200 copies/mL after 24 weeks of antiviral therapy or after scheme change.
* Informed consent signature

Exclusion Criteria:

* Younger than 18 years old.
* No virologic failure or RNA of VIH > 200 copies/mL.
* Presence of a serious opportunistic infection.
* Renal failure (including litiasis) or presence of gout.
* Pregnancy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2019-02-28 (Actual); Primary Completion 2020-03-30 (Estimated); Study Completion 2020-06-30 (Estimated)

PRIMARY OUTCOMES:
Viral load | Change from Baseline viral load at 3 months
  Number of viral copies/mL

SECONDARY OUTCOMES:
CD4+ count | Change from Baseline CD4+ count at 3 months
  Number of CD4+ cells

CONTACTS AND LOCATIONS:
Overall Officials: Enrique Teran, MD, PhD, Study Director — Universidad San Francisco de Quito
Locations (1):
- Hospital Enrique Garces, Quito, Ecuador

IPD SHARING:
Plan to Share IPD: Undecided